CLINICAL TRIAL: NCT00735800
Title: Psychosocial Telephone Intervention for Dementia Caregivers
Brief Title: Telephone Support for Dementia Caregivers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Geoffrey Tremont, Director, Neuropsychology, Rhode Island Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: R01NR010559 (NIH); R01NR010559 (NIH)
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Dementia
Keywords: Dementia; Caregivers; Alzheimer's disease
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supportive Counseling (Active Comparator)
  Interventions: Behavioral: Telephone Support
- Problem-Solving (Experimental)
  Interventions: Behavioral: Family Intervention:Telephone Tracking Support- Caregiver

INTERVENTIONS:
Behavioral: Family Intervention:Telephone Tracking Support- Caregiver — Family-based problem solving treatment
  Other Names: FITT-C
  Arms: Problem-Solving
Behavioral: Telephone Support — Supportive telephone counseling about caregiving
  Arms: Supportive Counseling

SUMMARY:
Caring for a patient with dementia is associated with increased feelings of burden and depression. The proposed study will examine the efficacy of Family Intervention: Telephone Tracking - Dementia (FITT-Dementia), a multi-component, family-based, telephone intervention, as a tool to reduce caregiver stress.

DETAILED DESCRIPTION:
A previous pilot study of this approach showed reduced burden and reaction to memory and behavior problems for dementia caregivers. This study will test the intervention in a larger group of caregivers and have a more detailed analysis of outcomes.

The caregiver of a person with dementia will receive telephone support calls. They will receive telephone calls from a trained member of the research team. These calls will occur over a six-month period and will be scheduled at a time that is convenient for the caregiver. They will receive a total of 16 calls over 6 months. During each call, the support person will discuss their current caregiving situation and provide various forms of support.

ELIGIBILITY:
Inclusion Criteria:

* 1) Diagnosis of dementia;
* 2) mild to moderate dementia;
* 3) family member or other adult in caregiver role for at least 6 months, and who provides at least 4 hours of supervision or direct assistance per day for the person with dementia;
* 4) care recipient lives in the community, including senior/retirement centers, but excluding nursing homes and assisted living centers; and
* 5) there is no plan for the care recipient to be placed in long term care or the caregiver to end their role within the next 6 months

Exclusion Criteria:

Patient:

* 1) other major medical condition affecting independent functioning
* 2) older than age 90; and
* 3) younger than age 50.

Caregiver:

* 1) major acute medical illness;
* 2) English not primary language;
* 3) cognitive impairment;
* 4) no access to a telephone; or
* 5) older than age 90.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2008-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Depression, burden, reaction to memory and behavior problems | Every two months, over a 6 month time-period , and a three month follow-up

SECONDARY OUTCOMES:
Cost-effectiveness and resource use | Monthly resource check-ins.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffery Tremont, Ph.D, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Background] Bruce JM, McQuiggan M, Williams V, Westervelt H, Tremont G. Burden among spousal and child caregivers of patients with mild cognitive impairment. Dement Geriatr Cogn Disord. 2008;25(4):385-90. doi: 10.1159/000122587. Epub 2008 Mar 29. PMID 18376128
- [Background] Davis JD, Tremont G. Impact of frontal systems behavioral functioning in dementia on caregiver burden. J Neuropsychiatry Clin Neurosci. 2007 Winter;19(1):43-9. doi: 10.1176/jnp.2007.19.1.43. PMID 17308226
- [Background] Epstein-Lubow G, Davis JD, Miller IW, Tremont G. Persisting burden predicts depressive symptoms in dementia caregivers. J Geriatr Psychiatry Neurol. 2008 Sep;21(3):198-203. doi: 10.1177/0891988708320972. PMID 18838742
- [Background] Spitznagel MB, Tremont G, Davis JD, Foster SM. Psychosocial predictors of dementia caregiver desire to institutionalize: caregiver, care recipient, and family relationship factors. J Geriatr Psychiatry Neurol. 2006 Mar;19(1):16-20. doi: 10.1177/0891988705284713. PMID 16449755
- [Background] Steadman PL, Tremont G, Davis JD. Premorbid relationship satisfaction and caregiver burden in dementia caregivers. J Geriatr Psychiatry Neurol. 2007 Jun;20(2):115-9. doi: 10.1177/0891988706298624. PMID 17548782
- [Background] Tremont G, Davis JD, Bishop DS. Unique contribution of family functioning in caregivers of patients with mild to moderate dementia. Dement Geriatr Cogn Disord. 2006;21(3):170-4. doi: 10.1159/000090699. Epub 2006 Jan 3. PMID 16397397
- [Background] Tremont G, Davis JD, Bishop DS, Fortinsky RH. Telephone-Delivered Psychosocial Intervention Reduces Burden in Dementia Caregivers. Dementia (London). 2008;7(4):503-520. doi: 10.1177/1471301208096632. PMID 20228893
- See also: Link to study webpage — http://www.rhodeislandhospital.org/rih/services/alzheimers/Dementia.htm